CLINICAL TRIAL: NCT06133946
Title: Cohort of Universal Newborn Deafness-gene Screening in Nantong City, China
Brief Title: Cohort Of DEafness-gene Screening
Acronym: CODES
Status: Active, not recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Nantong Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Gang Qin, MD, PhD, Associate Professor, Affiliated Hospital of Nantong University
Other Study IDs: BE2015655
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss
Keywords: Newborn hearing screening; Genetic screening; Cohort study
MeSH Terms: conditions — Hearing Loss | interventions — Genetic Testing; Otoacoustic Emissions, Spontaneous; Evoked Potentials, Auditory, Brain Stem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spot specimen was collected from the infants' heel sticks. Genomic DNA was extracted by a blood filter paper nucleic acid extraction kit (CapitalBio, Beijing, China) and tested using a deafness gene variant detection array kit (CapitalBio, Beijing, China) with LuxScan 10K-B Microarray Scanner (CapitalBio, Beijing, China).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined screening: All newborns underwent combined hearing and genetic screening.
  Interventions: Genetic: Genetic screening test (Deafness gene variant detection array kit)

INTERVENTIONS:
Genetic: Genetic screening test (Deafness gene variant detection array kit) — Infant participants were screened for fifteen variants in four genes (i.e., GJB2, SLC26A4, MT-RNR1 and GJB3).
  Other Names: Newborn hearing screening test (otoacoustic emission, OAE); Hearing re-screening test (OAE and automated auditory brainstem response [AABR]）; Hearing diagnostic test (auditory brainstem response [ABR] and auditory steady state response [ASSR])

SUMMARY:
This study was based on a concurrent newborn genetic and hearing screening program in Nantong city. From January 2016 to December 2020, newborn infants were recruited and received combined screening for free, funded in part by the municipal government and research project foundations. The population-based longitudinal databank for all children with hearing loss in Nantong city commenced in January 2016 and maintained indefinite recruitment and ongoing follow-up.

DETAILED DESCRIPTION:
The severity of hearing loss was graded as mild (26-40 dB), moderate (41-60 dB), severe (61-80 dB), and profound (≥81 dB).

Genomic DNA was extracted by a blood filter paper nucleic acid extraction kit (CapitalBio, Beijing, China) and tested using a deafness gene variant detection array kit (CapitalBio, Beijing, China) with LuxScan 10K-B Microarray Scanner (CapitalBio, Beijing, China). The genetic screening entailed genotyping 15 variants in 4 genes: c.35delG, c.176_191del16, c.235delC, c.299_300delAT (GJB2 gene); c.1174A>T, c.1226G>A, c.1229C>T, c.1975G>C, c.2027T>A, c.2168A>G, c.IVS7-2A>G, c.IVS15 + 5G>A (SLC26A4 gene); m.1494C>T, m.1555A>G (MT-RNR1 gene); c.538C>T (GJB3 gene). The results were categorized as (1) negative, (2) carrier (GJB2 or SLC26A4, heterozygous mutations; MT-RNR1 mutations; GJB3 mutations; or heterozygous mutations in multiple genes), and (3) refer (GJB2 or SLC26A4, homozygous or compound heterozygous mutations).

This study was approved by the ethics committees of Nantong municipal Health Commission and all hospitals involved. Written informed consent was obtained from the infant's parents.

This study followed the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) reporting guideline for cohort studies.

ELIGIBILITY:
Inclusion Criteria:

1. The infants were born between January 2016 and December 2020;
2. The infants' health condition was good enough to tolerate the screening procedures;
3. The parents were urban residents of Nantong city;
4. The parents agreed to have their babies participating in the combined hearing and genetic screening program.

Exclusion Criteria:

1. The infants' blood samples were unqualified for the genetic tests according to criteria of the National Health Commission of China's technical specification for neonatal screening of congenital diseases;
2. The infants were lost to follow-up.

Ages: 3 Days to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants were newborn infants born between January 2016 and December 2020 from the Han population in Nantong city, China.
Sampling Method: Non-Probability Sample
Enrollment: 35920 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of hearing loss at age of 3 months | From Jan 1, 2016 to Mar 31, 2021
  Diagnosis of HL was confirmed by hearing diagnostic tests (ABR+ASSR) at age of 3 months.
  Auditory steady-state response (ASSR) were used as an alternative and adjunct to the auditory brainstem response (ABR) for threshold estimation.

SECONDARY OUTCOMES:
Language ability of HL children at ages of 5 years and 8 years | From Jan 1, 2021 to Dec 31, 2028
  Mandarin sentence repetition task (MSRT) was used to reflect the children's language ability.
Receptive vocabulary of HL children at ages of 5 years and 8 years | From Jan 1, 2021 to Dec 31, 2028
  The Chinese version of the Peabody Picture Vocabulary Test-Revised (C-PPVT-R, Lu & Liu, 1998) was used to evaluate children's expressive vocabulary ability. The possible score ranged from 0-125, and test-retest reliability was exceeded 0.9.
Non-verbal IQ of HL children at ages of 5 years and 8 years | From Jan 1, 2021 to Dec 31, 2028
  The Chinese version of the Test of Nonverbal Intelligence, fourth edition (C-TONI-4, Lin et al., 2016) was used to evaluate children's nonverbal intelligence regarding problem solving and abstract reasoning. The possible score ranged from 0 to 48, and internal consistency reliability was 0.87.

IPD SHARING:
Plan to Share IPD: No